CLINICAL TRIAL: NCT03918512
Title: Development and Validation of a Questionnaire for Assessing Activity Limitation in Patients With Lumbar Spinal Stenosis : The Cochin L3S Questionnaire.
Acronym: CL3S
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180412
Record Dates: First submitted 2019-03-15; First posted 2019-04-17 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar spinal stenosis; LSS specific activity limitation; development and validation of new questionaire
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: nine online self-administered questionnaires — patients will be invited to complete the following nine online self-administered questionnaires at baseline, 7 days and 3 months:
  * Demographical and clinical characteristics at baseline
  * Consolidated version of the CSS-48 questionnaire
  * Lumbar pain numeric rating scale (NRS)
  * Radicular pain NRS
  * Zurich Claudication Questionnaire (ZCQ) (physical function subscale)
  * Oswestry Disability Index (ODI)
  * Fukushima LSS Scale 25 (FLS-25)
  * 12-Item Short Form Health Survey (SF-12)
  * Anchoring questions : 1 anchoring question about patient acceptable symptom state (at baseline, 7 days and 3 month) and 1 anchoring question about patient minimal clinically important difference (at 3 months).

SUMMARY:
To develop and validate a questionnaire aiming at assessing specific activity limitation in patients with lumbar spinal stenosis (LSS).

DETAILED DESCRIPTION:
Construction of the provisional questionnaire :

In a first step, semi-structured in-depth individual interviews were conducted from September 20, 2016 to January 4, 2017, in 20 patients fulfilling inclusion criteria to collect concepts related to LSS-specific activity limitation, participation restriction and patients' views about their condition. Thematic content was analysed using investigator triangulation. Overall, 57 items were generated by patients. 48 items were related to LSS-specific activity limitation and were used to construct the provisional 48-item Cochin L3S questionnaire (CL3S-48). Acceptability and understandability of the provisional CL3S-48 questionnaire was tested and consolidated in 10 patients with LSS.

Item reduction and validation of the questionnaire :

In a second step, 200 eligible patients according to our medical records will be informed by email of the purpose of the study, their non-opposition to the collection of data will be collected and patients will be invited to complete the following online self-administered questionnaires at baseline, 7 days and 3 months:

* Demographical and clinical characteristics at baseline
* Consolidated version of the CL3S-48 questionnaire
* Lumbar pain numeric rating scale (NRS)
* Radicular pain NRS
* Zurich Claudication Questionnaire (ZCQ) physical function subscale
* Oswestry Disability Index (ODI)
* Fukushima LSS Scale 25 (FLS-25)
* 12-Item Short Form Health Survey (SF-12)
* 1 anchoring question about patient acceptable symptom state
* 1 anchoring question about patient minimal clinically important difference at 3 months.

In a third step, the number of items will be reduced according to their metrological qualities. The psychometric properties of the new scale will be assessed and the scale will be consolidated to provide the final questionnaire

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 50 year old
* with lumbar spinal stenosis (LSS) according to medical records.

Exclusion Criteria:

* lumbar spinal surgery,
* cognitive impairment and inability to speak and/or understand French.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatology Department of Limoges Hospital and the Rehabilitation Department of Cochin Hospital, Paris
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Lumbar Spinal Stenosis-specific activity limitation in patients with Lumbar Spinal Stenosis | at baseline
  To develop and validate a questionnaire aiming at assessing specific activity limitation in patients with LSS

CONTACTS AND LOCATIONS:
Overall Officials: Christelle NGUYEN, MD, PhD, Principal Investigator — APHP (assistance publique hôpitaux de Paris)
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No